CLINICAL TRIAL: NCT03073356
Title: Effects of Ketones on Cardiac Function and Oxygen Consumption in Heart Failure Patients With Reduced Ejection Fraction and Healthy Test Subjects
Brief Title: Ketones in Heart Failure - Effects on Cardiac Efficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-10-72-316-16
Record Dates: First submitted 2017-02-20; First posted 2017-03-08 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-01

CONDITIONS: Heart Failure, Systolic; Ketonemia
Keywords: Myocardial metabolism; Positron emission tomography; Echocardiography; Right sided heart catheterization
MeSH Terms: conditions — Heart Failure, Systolic; Ketosis

STUDY DESIGN:
Intervention Model Description: Randomized dobbel-blinded crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control - Healthy test subjects (Experimental): Age matched subjects without symptoms of heart failure or ischemic heart disease N=10
  Interventions: Biological: Infusion of 3-OHB; Biological: Infusion of placebo
- HFrEF - Heart failure patients investigated by PET (Experimental): Patients with heart failure (HFrEF) N=12
  Interventions: Biological: Infusion of 3-OHB; Biological: Infusion of placebo
- HFrEF - Right heart catheterization (Experimental): Patients with heart failure (HFrEF) N=12
  Interventions: Biological: Infusion of 3-OHB; Biological: Infusion of placebo
- HFrEF - Right heart catheterization study 2 (Experimental): Dose finding study (increasing dosage of 3-OHB)
  Interventions: Biological: Infusion of 3-OHB; Biological: Infusion of placebo

INTERVENTIONS:
Biological: Infusion of 3-OHB — Increase in 3-OHB levels
  Other Names: Na-3-OHB
Biological: Infusion of placebo — NaCl
  Other Names: NaCl

SUMMARY:
Ketones may have beneficial effects on myocardial metabolism and hemodynamics. In the present study, healthy test subjects and patients with heart failure with reduced ejections fraction will be investigated in a randomized cross-over design with ketone infusions and placebo. Myocardial efficiency and hemodynamics will be evaluated.

DETAILED DESCRIPTION:
The prevalence of patients with heart failure and reduced ejection fraction (HFrEF) is 1-2%, and the lifetime risk of heart failure at age 55 years is approximately 30%. Despite advances in treatment, hospitalization rate and mortality remains high. It is well known that myocardial metabolism changes during development of HFrEF, and may contribute to contractile dysfunction. However, the myocardium can be considered an omnivore regarding substrate utilization, conferring an important adaptive property. Hence, it metabolizes either glucose, lipids, lactate, amino acids or ketones (3-hydroxybutyrate) depending on substrate availability, hormonal status and cardiac demands. These substrates differ with regard to myocardial energy efficiency (MEE) (cardiac work related to oxygen consumption). Since high MEE is associated with a better prognosis in HFrEF, manipulating substrate uptake could be a new treatment modality in heart failure patients.

Recently, it was shown that the human myocardium increases 3-hydroxybutyrate (3-OHB) metabolism during development of HFrEF. These changes may be beneficial as 3-OHB could increase myocardial efficiency and lower oxidative stress by scavenging free radicals. However, until now this has not been investigated in clinical trials, and the effect of 3-OHB on cardiac function, oxygen consumption and perfusion remains undetermined in HFrEF patients.

In the present study the investigators will evaluate whether elevated circulating 3-OHB affect myocardial oxygen consumption, MEE and perfusion in healthy subjects and patients with HFrEF, and whether 3-OHB affect hemodynamics and contractile function.

10 healthy test subjects and 20 HFrEF patients will be subjected to placebo and 3-OHB infusion in a randomized cross-over design. Acetate-PET, echocardiography and right sided heart catheterization will be applied.

ELIGIBILITY:
Inclusion Criteria:

* For participants with heart failure:
* Symptoms of Heart failure NYHA 2-3
* LVEF<40%

For all participants:

* Negative HCG for women in the pregnant age

Exclusion Criteria:

* Significant cardiac valve disease
* Signs or history of major myocardial infarction (STEMI) within 3 months
* Other disease or treatment making subject unsuitable for study participation
* Treatment for diabetes or HbA1c level >7%

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Myocardial efficiency | 1 day
  Based on myocardial PET examinations
Cardiac output | 1 day
  Right sided heart catheterization

SECONDARY OUTCOMES:
Myocardial perfusion | 1 day
  Based on myocardial PET examinations
Myocardial oxygen consumption | 1 day
  Based on myocardial PET examinations
Pulmonary and wedge pressure | 1 day
  Right sided heart catheterization
Mixed venous saturation | 1 day
  Right sided heart catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Roni R Nielsen, MD PHD, Principal Investigator — Dept. of Cardiology
Locations (1):
- Dept. of cardiology, Aarhus university hospital Skejby, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No